CLINICAL TRIAL: NCT06735989
Title: Effects of a Moral Reasoning Intervention on Moral Justification Abilities
Brief Title: Moral Reasoning Intervention on Moral Justification Abilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Prof., IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Moral-REA
Record Dates: First submitted 2024-07-31; First posted 2024-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Moral Development; Moral Dilemma; Healthy Controls; Moral Justification

STUDY DESIGN:
Intervention Model Description: Intervention study, monocentric, randomized, double-blind, and multiparametric.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be maintained for allocation concealment, which will be carried out through closed and opaque mails by a blind operator. Subjects will be labelled with a numerical code to ensure anonymisation. Subjects, teachers, evaluators and statisticians will be blind to allocation. Specifically, teachers of both groups will be not informed about the aim of the study. They will be provided with specular material for the seminar (same structure and number of slides). They will be only informed to not answer to specific questions about dilemmas. Subjects of a group will be informed that the other group is attending a seminar on "reasoning". They will be separated until the end of the post-test phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moral (Experimental): The Moral group will read a short text explaining the meaning and function of moral justification, and outlining brief descriptions of six morally relevant factors. The Moral group will then attend a 1h30 lecture on moral reasoning.
  Interventions: Other: Lecture on moral reasoning
- Non-moral (Active Comparator): The Non-moral will read a short text explaining the meaning and function of argumentation, and outlining brief descriptions of six logical and argumentative principles. The Non-moral group will then attend a 1h30 lecture on (non-moral) logical reasoning.
  Interventions: Other: Lecture on logical reasoning

INTERVENTIONS:
Other: Lecture on moral reasoning — One and a half-hour long lecture on moral justification and moral reasoning
  Arms: Moral
Other: Lecture on logical reasoning — One and a half-hour long lecture on logical and argumentative principles
  Arms: Non-moral

SUMMARY:
The primary aim of this study is to evaluate the short (immediate) and mid-term (one month) impact of moral (vs non-moral) reasoning interventions on the moral justification abilities in non-expert subjects. Such an impact will be assessed by observing quantitative changes (on 1 to 4 points scale) of qualitative variables in the moral justification expressed by the subjects.

DETAILED DESCRIPTION:
The aim of this study is to test wether a single intervention on moral reasoning can have short and/or mid-term effects on the justification of moral judgements about a problematic moral case. Focusing on justification allows to assess reasonable improvement by referring to a procedural standard, that is, without assuming any substantive normative view; namely, without evaluating a "betterment" on the basis of the content of moral judgements, but rather on the satisfaction of formal, procedural conditions in their justification. Our standard for a good moral justification consists in a set of procedural features, such as logical, empirical, and conceptual competence, openness to revision, sympathetic imagination, and bias avoidance.

Once enrolled, participants will be randomized through random.org software in the two experimental groups: 1) the moral and 2) the non-moral condition. Allocation concealment will be carried out through closed and opaque mails by a blind operator. Subjects will undergo a neuropsychological assessment and a (optional) task-based fMRI at study entry. Furthermore, during the day of the intervention (seminar: moral or logical reasoning), participants will undergo a pre-test (before the intervention) and a post-test (after the intervention) on a morally problematic case. The same test will be repeated by all participants one month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* University students (other than Philosophy) within the first 3 years
* Aged between 18 and 26 years old
* Italian speakers
* Oral and written informed consent to study participation

Exclusion Criteria:

* A current psychiatric condition
* Contraindications to MRI study (cardiac pacemakers; metal splinters or fragments; metal protheses not compatible with the magnetic field; claustrophobia; women who are pregnant or intending to become pregnant during the study; breastfeeding women).

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Short and mid-term (one month) impact of moral vs non-moral reasoning interventions on moral justification abilities in non-expert subjects when performing a moral dilemma. | Baseline, 5 weeks
  The primary aim of this study is to evaluate the short (immediate) and mid-term (one month) impact of moral (vs non-moral) reasoning interventions on the moral justification abilities in non-expert subjects. Such an impact will be assessed by observing quantitative changes (on a 0 to 3 points scale) in the moral justifications expressed by the subjects in six domains: empirical competence, conceptual competence, logical coherence, sympathetic imagination, bias reduction, openness to revision of opinions.

SECONDARY OUTCOMES:
Relationship between brain BOLD activity during task-based fMRI and changes in moral justification abilities. | Baseline, 5 weeks
  To investigate the relationship between pre-intervention subjects' brain BOLD activity during a task-based functional MRI (fMRI), using a moral reasoning paradigm, and changes in moral justification abilities in six domains (empirical competence, conceptual competence, logical coherence, sympathetic imagination, bias reduction, openness to revision of opinions) assessed using a 0-3 point scale.
Relationship between brain BOLD activity during task-based fMRI and agreement with moral statements. | Baseline, 5 weeks
  To investigate the relationship between pre-intervention subjects' brain BOLD activity during a task-based functional MRI (fMRI), using a moral reasoning paradigm, and agreement with moral statements assessed using a 0-3 point scale.
Relationship between brain BOLD activity during task-based fMRI and confidence post-intervention. | Baseline, 5 weeks
  To investigate the relationship between pre-intervention subjects' brain BOLD activity during a task-based functional MRI (fMRI), using a moral reasoning paradigm, and confidence post-intervention assessed by using 0-3 point scales.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

REFERENCES:
- [Background] Greene JD. The rat-a-gorical imperative: Moral intuition and the limits of affective learning. Cognition. 2017 Oct;167:66-77. doi: 10.1016/j.cognition.2017.03.004. Epub 2017 Mar 23. PMID 28343626
- [Background] Greene JD, Sommerville RB, Nystrom LE, Darley JM, Cohen JD. An fMRI investigation of emotional engagement in moral judgment. Science. 2001 Sep 14;293(5537):2105-8. doi: 10.1126/science.1062872. PMID 11557895
- [Background] Haidt J. The emotional dog and its rational tail: a social intuitionist approach to moral judgment. Psychol Rev. 2001 Oct;108(4):814-34. doi: 10.1037/0033-295x.108.4.814. PMID 11699120
- [Background] Kahneman D, Klein G. Conditions for intuitive expertise: a failure to disagree. Am Psychol. 2009 Sep;64(6):515-26. doi: 10.1037/a0016755. PMID 19739881
- [Background] Klenk M, Sauer H. Moral Judgement and Moral Progress: The Problem of Cognitive Control. Philos Psychol. 2021 Jul 2;34(7):938-961. doi: 10.1080/09515089.2021.1931670. eCollection 2021. PMID 34556899
- [Background] Rozin P, Haidt J, Fincher K. Psychology. From oral to moral. Science. 2009 Feb 27;323(5918):1179-80. doi: 10.1126/science.1170492. No abstract available. PMID 19251619
- [Background] Schaefer GO, Savulescu J. Procedural Moral Enhancement. Neuroethics. 2019;12(1):73-84. doi: 10.1007/s12152-016-9258-7. Epub 2016 Apr 20. PMID 30956726
- [Background] Schwitzgebel E, Cokelet B, Singer P. Do ethics classes influence student behavior? Case study: Teaching the ethics of eating meat. Cognition. 2020 Oct;203:104397. doi: 10.1016/j.cognition.2020.104397. Epub 2020 Jul 25. PMID 32721655
- [Background] Schwitzgebel E, Cushman F. Philosophers' biased judgments persist despite training, expertise and reflection. Cognition. 2015 Aug;141:127-37. doi: 10.1016/j.cognition.2015.04.015. Epub 2015 May 14. PMID 25981733